CLINICAL TRIAL: NCT01184638
Title: Long-term Outcome Followed-up of the Cognitive Disorders After General Anesthesia
Brief Title: Long-term Outcome of General Anesthesia on Dysgnosia
Acronym: LOGAND
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Fu Zhou Wang, Dr, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NJMU-2010-07022; NJFY7M12
Record Dates: First submitted 2010-08-16; First posted 2010-08-19 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Delirium,; Dementia,; Amnestic,; Cognitive Disorders
Keywords: Cognitive Disorders; General anesthesia; Sevoflurane; Propofol; Memory
MeSH Terms: conditions — Delirium; Dementia; Cognitive Dysfunction | interventions — Sevoflurane; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Local anesthesia (No Intervention): Patients received local anesthesia without any intervention of general anesthetics
- Inhalational anesthesia (Active Comparator): Patients received sevoflurane anesthesia during general anesthesia
  Interventions: Drug: Sevoflurane
- Intravenous anesthesia (Active Comparator): Patients received intravenous anesthetic (Propofol) during general anesthesia
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Sevoflurane — 1-8% sevoflurane for maintaining the whole period of general anesthesia
  Other Names: Sevorane
  Arms: Inhalational anesthesia
Drug: Propofol — 1-4 mg/kg/h of propofol during the whole period of general anesthesia
  Other Names: Diprivan
  Arms: Intravenous anesthesia

SUMMARY:
Cognitive disorders in patients underwent general anesthesia are discussed for decades, but whether there were precise relationship between general anesthesia and dysgnosia is yet to be guaranteed. Although controversial data reported from experimental studies in animals, the investigators still proposed that general anesthetics could impair the normally organized system of the central nervous system, which finally displayed a dysfunction of cognition after general anesthesia in a short- or long-term period. Therefore, different types of general anesthetics such as inhalational anesthetics and intravenous anesthetics, the investigators hypothesized, had a long-term influence on patients' cognitive ability.

ELIGIBILITY:
Inclusion Criteria:

* Patients with informed consents
* Without basal disorders of neurology and psychiatrics

Exclusion Criteria:

* With the history of cognitive disorders
* With chronic neurological disorders
* Cannot communicate with investigators
* Cannot stand general anesthesia

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2010-08; Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Cognitive ability | The 10th year since postoperation
  Cognitive ability will be assessed with digital lignature game, figure identificaiton, and recall memory

SECONDARY OUTCOMES:
Cognitive ability | One hour before operation
  Cognitive ability will be assessed with digital lignature game, figure identificaiton, and recall memory
Cognitive ability | Immediately after operation (0 day)
  Cognitive ability will be assessed with digital lignature game, figure identificaiton, and recall memory
Cognitive ability | One month after operation
  Cognitive ability will be assessed with digital lignature game, figure identificaiton, and recall memory
Cognitive ability | Six month after operation
  Cognitive ability will be assessed with digital lignature game, figure identificaiton, and recall memory
Cognitive ability | One year after operation
  Cognitive ability will be assessed with digital lignature game, figure identificaiton, and recall memory
Cognitive ability | Once a year from the 1st year after operation up to 9th year
  Cognitive ability will be assessed with digital lignature game, figure identificaiton, and recall memory

CONTACTS AND LOCATIONS:
Overall Officials: FuZhou Wang, PhD MD, Study Director — Nanjing Medical University
Locations (1):
- Nanjing Maternity and Child Health Care Hospital, Nanjing, Jiangsu, China